CLINICAL TRIAL: NCT06514144
Title: Exacerbations and Real-World Outcomes Among Chronic Obstructive Pulmonary Disease Patients Receiving Breztri (EROS Study)
Brief Title: Exacerbations Among Patients Receiving Breztri (EROS Study)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00079
Record Dates: First submitted 2024-03-18; First posted 2024-07-23 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Disease; Chronic Obstructive; Retrospective Studies
Keywords: COPD; Delayed therapy; Exacerbations; Triple therapy
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Treatment Initiation: Initiation of treatment following exacerbation classified as prompt, delayed or very delayed.
  Interventions: Drug: BGF

INTERVENTIONS:
Drug: BGF — budesonide/glycopyrrolate/formoterol fumarate
  Other Names: Breztri

SUMMARY:
EROS was a retrospective analysis of people with COPD using the MORE2 Registry®. Inclusion required ≥1 severe, ≥2 moderate, or ≥1 moderate exacerbation while on other maintenance treatment. Primary outcomes were the rate of COPD exacerbations and healthcare costs for those that received BGF promptly. The effect of each 30-day delay in initiation of BGF was estimated using a multivariable negative binomial regression model.

DETAILED DESCRIPTION:
EROS was a retrospective real-world evidence claims analysis study, assessing the relationship between the timing of Breztri Aerosphere following an exacerbation and the appearance of subsequent disease exacerbations of people with COPD.

The study used administrative claims data in the US sourced from the Inovalon MORE2 Registry® between July 2019 and March 2022. Inclusion required one of the following qualifying exacerbation events: ≥1 severe, ≥2 moderate, or ≥1 moderate exacerbation while on other maintenance treatment, be age ≥40 at the index date, and have ≥90 days of continuous enrollment following the index date.

Primary outcomes were the rate of COPD exacerbations and healthcare costs for those that received BGF promptly. The effect of each 30-day delay in initiation of BGF was estimated using a multivariable negative binomial regression model. Statistical analyses included both descriptive and multivariable approaches- negative binomial regression models to estimate the effect of each 30-day delay on the number of exacerbations and a gamma model with a log-link to estimate the effects on the incremental increase in COPD-related costs.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 1 prescription fill for BGF on or following July 24th, 2020 (Breztri approval date);
* Evidence of any of the following exacerbation patterns within the 12-month period preceding the initiation of BGF, all index exacerbation events must occur following BGF approval: (1) one moderate exacerbation (the exacerbation must occur following approval of Breztri) with presence of other inhaled therapy, (2) two moderate exacerbations (the second exacerbation must occur following approval of Breztri) without the presence of other inhaled therapy, or (3) Severe Exacerbation- Inpatient COPD hospitalization
* ≥ 12 months of continuous enrollment preceding the index exacerbation date
* ≥ 90 days of continuous enrollment following the index exacerbation date
* Age ≥ 40 years on the index exacerbation date

Exclusion Criteria:

* Presence of closed triple therapy during the baseline period
* Initiation of BGF 4/1/2022 or later
* Presence of an enrollment gap of more than 14-days from index exacerbation date to BGF initiation date

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with COPD who experienced a COPD exacerbation event and were subsequently initiated on therapy with budesonide/glycopyrrolate/formoterol fumarate (BGF); sourced from secondary administrative claims data between July 2020 through March 2022.
Sampling Method: Non-Probability Sample
Enrollment: 2409 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
COPD Exacerbation events | Annualized rates from index exacerbation through end of data availability, an average follow-up time of 331 days.
  Annualized rates of COPD exacerbation events observed from index date (qualifying exacerbation event) through study completion (until end of data availability), an average follow-up time of 331 days.

SECONDARY OUTCOMES:
Healthcare resource utilization | Annualized rates from index exacerbation through end of data availability, an average follow-up time of 331 days.
  Annualized rates of health care services observed (e.g., inpatient visits, ER visits) from index date (qualifying exacerbation event) through study completion (until end of data availability), an average follow-up time of 331 days.
Healthcare costs | Annualized costs from idex exacerbation through end of data availability, an average follow-up time of 331 days.
  Annualized costs of health care services observed (e.g., total health care costs, total-COPD related costs) from index date (qualifying exacerbation event) through study completion (until end of data availability), an average follow-up time of 331 days.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pollack, MS, Study Director — AstraZeneca
Locations (1):
- AstraZeneca, Wilmington, Delaware, United States

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5980R00079&attachmentIdentifier=ed83ff39-7b76-4b7c-9791-166c16f2664e&fileName=EROS_(D5980R00079)_CSR_Synopsis_Redacted2.pdf&versionIdentifier=